CLINICAL TRIAL: NCT06952400
Title: T1622 The Registry Study of Genetic Alterations of Melanoma in Taiwan
Brief Title: The Registry Study of Genetic Alterations of Melanoma in Taiwan
Acronym: Melanoma
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T1622
Record Dates: First submitted 2025-04-06; First posted 2025-04-30 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Primary Melanoma of the Extremity
Keywords: next-generation sequencing; acral melanoma; mucosal melanoma; cutaeous melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor Sample(s):
  One H&E staining slide, and 10 tissue slides for cancer panel-based next generation sequencing analysis, including fusion panel will be required (first priority).
  The other one H&E staining slide and 5 slides (4-5 um thickness) will be lab for RNA extraction (optional, operative tissue was favored). IHC for possible biomarkers (including MDM2/HER2): one H&E staining slide and 5 slides.
  Non-tumor Sample (Blood): Fifteen (15) ml of blood will be collected from the participant: 7 ml in EDTA tube (purple top) and 8 ml in Cell-Free DNA blood collection tube.
  Non-tumor Sample (Stool for microbiota): Fecal sample preparation and sequencing will be performed at CGMH. 16S rRNA gene sequencing will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: (early acral melanoma): melanoma stage I/II
- Cohort 2: (locally advanced acral melanoma): melanoma, stage III, resectable
- Cohort 3: (advanced): unresectable / metastatic melanoma, stage III/IV or recurrent melanoma (unresectable). Staging is based on AJCC Cancer Staging System 8th edition).
- Cohort 4: The patients with advanced melanoma with available comprehensive NGS report are included in cohort

SUMMARY:
Cutaneous melanoma is the most aggressive malignancy in skin cancers. Cutaneous melanoma is a rare disease in Taiwan with an incidence rate of around 1/100,000. Acral lentiginous melanoma is the most common subtype and comprises more than half of cutaneous melanoma in Asia including Taiwan but only 1% in Caucasians. In addition, mucosal melanoma accounts for more than 20% of malignancy melanoma in Taiwan but only 1% in Caucasians. Acral and mucosal melanomas have distinct epidemiological, clinical, pathological and genetic features from non-acral melanoma which is commonly seen in Western countries. Comparing with melanoma in Caucasians, Asian melanoma has higher recurrence rate after primary surgery, lower response rate to immunotherapy, and shorter progression-free survival for immunotherapy and targeted therapy leading generally poor survival outcomes regardless stage.

DETAILED DESCRIPTION:
Most melanoma patients present with locally advanced or metastatic disease at diagnosis reflecting the aggressive disease nature of melanoma in Taiwan. Currently, surgical resection of primary tumor and lymph node dissection are the main treatment for patients with locally advanced melanoma. Adjuvant therapy should be considered for stage III melanoma. Unfortunately, most patients recur after above aggressive treatment. Systemic treatment including targeted therapy, immunotherapy and chemotherapy is the main for unresectable or metastatic melanoma. The prognosis of these patients remains poor with a median survival time around a year. Therefore, a better understanding of this deadly disease is crucial and finding better therapeutic strategies for these patients and stratifying patients with suitable treatment are urgent.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Pathologically confirmed melanoma. (Patients with additional malignancies requiring treatment or follow-up are allowed. Only treatment for melanoma should be recorded).
3. ECOG performance status < 3
4. Cohort 1(early acral melanoma): melanoma, stage I/II; Cohort 2 (locally advanced acral melanoma): melanoma, stage III, resectable; and Cohort 3 (advanced): unresectable / metastatic melanoma, stage III/IV or recurrent melanoma (unresectable). Staging is based on AJCC Cancer Staging System 8th edition). The patients with advanced melanoma with available comprehensive NGS report are included in cohort 4.
5. Willingness to provide archival or newly obtained tumor tissues for this study proposal
6. Life expectancy more than 3 months -
7. Patients fully understand the protocol with the willingness to have regular follow-up

Exclusion Criteria:

1. Inability to cooperate by providing a complete medical history
2. No available tumor tissues for genetic testing (archived tissue sampling more than 5 years from screening date)
3. Undesirable compliance (Mental status is not fit for further treatment or data collection.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1(early acral melanoma): melanoma, stage I/II; Cohort 2 (locally advanced acral melanoma): melanoma, stage III, resectable; and Cohort 3 (advanced): unresectable / metastatic melanoma, stage III/IV or recurrent melanoma (unresectable). Staging is based on AJCC Cancer Staging System 8th edition). The patients with advanced melanoma with available comprehensive NGS report are included in cohort 4.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the evolution of acral melanoma patients in Taiwan. | Duration of Enrollment: 2022/10-2025/12
  1. Collecting the tissues from melanoma patients for NGS studies, One H&E staining slide, and 10 tissue slides (4-5 um thickness) for cancer panel-based next generation sequencing analysis, including fusion panel (10 slides) will be required (first priority).
  2. Non-tumor Sample (Blood): Fifteen (15) ml of blood will be collected from the participant: 7 ml in EDTA tube (purple top) and 8 ml in Cell-Free DNA blood collection tube. These blood samples will be separated into peripheral blood mononuclear cells and plasma specimens for germline mutation analysis and potential biomarker study, respectively.
  3. Non-tumor Sample (Stool for microbiota):Collecting stool specimens before systemic treatment (for prospective cohort), 2-3 months after initiating targeted therapy or immunotherapy. IHC staining for specific biomarkers such as MDM2 and HER2 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Chiao-En Wu, MD, PhD, Principal Investigator — Chang Gung Medical Foundation; Tsang-Wu Liu, MD, Study Chair — Taiwan Cooperative Oncology Group,National Health Research Institutes, Taiwan; Nai-Jung Chiang, MD, PhD, Principal Investigator — Taiwan Cooperative Oncology Group,National Health Research Institutes, Taiwan
Locations (16):
- Taiwan (16):
  - Taipei Veterans General Hospital, Taipei, Taiwan/Taipei
  - CHANG GUNG MEMORIAL HOSPITAL, Chiayi, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University, Kaohsiung City
  - National Taiwan University Hospital ,NTUH Hsin-Chu Branch, Sindian City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University -Ministry of Health and Welfare Shuang-Ho Hospital, Taipei
  - Wan Fang Hospital, Taipei Medical University, Taipei
  - CHANG GUNG MEMORIAL HOSPITAL, Linkou, Taoyuan District
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Result] Chang JW, Huang YL, Chang YY, Lo YF, Ho TY, Huang YT, Chen HW, Wu CE. Sentinel Lymph Node Biopsy Was Associated With Favorable Survival Outcomes For Patients With Clinically Node-Negative Asian Melanoma. Cancer Manag Res. 2019 Nov 14;11:9655-9664. doi: 10.2147/CMAR.S227837. eCollection 2019. PMID 31814762
- [Result] Hayward NK, Wilmott JS, Waddell N, Johansson PA, Field MA, Nones K, Patch AM, Kakavand H, Alexandrov LB, Burke H, Jakrot V, Kazakoff S, Holmes O, Leonard C, Sabarinathan R, Mularoni L, Wood S, Xu Q, Waddell N, Tembe V, Pupo GM, De Paoli-Iseppi R, Vilain RE, Shang P, Lau LMS, Dagg RA, Schramm SJ, Pritchard A, Dutton-Regester K, Newell F, Fitzgerald A, Shang CA, Grimmond SM, Pickett HA, Yang JY, Stretch JR, Behren A, Kefford RF, Hersey P, Long GV, Cebon J, Shackleton M, Spillane AJ, Saw RPM, Lopez-Bigas N, Pearson JV, Thompson JF, Scolyer RA, Mann GJ. Whole-genome landscapes of major melanoma subtypes. Nature. 2017 May 11;545(7653):175-180. doi: 10.1038/nature22071. Epub 2017 May 3. PMID 28467829
- [Result] Newell F, Wilmott JS, Johansson PA, Nones K, Addala V, Mukhopadhyay P, Broit N, Amato CM, Van Gulick R, Kazakoff SH, Patch AM, Koufariotis LT, Lakis V, Leonard C, Wood S, Holmes O, Xu Q, Lewis K, Medina T, Gonzalez R, Saw RPM, Spillane AJ, Stretch JR, Rawson RV, Ferguson PM, Dodds TJ, Thompson JF, Long GV, Levesque MP, Robinson WA, Pearson JV, Mann GJ, Scolyer RA, Waddell N, Hayward NK. Whole-genome sequencing of acral melanoma reveals genomic complexity and diversity. Nat Commun. 2020 Oct 16;11(1):5259. doi: 10.1038/s41467-020-18988-3. PMID 33067454
- [Result] Newell F, Kong Y, Wilmott JS, Johansson PA, Ferguson PM, Cui C, Li Z, Kazakoff SH, Burke H, Dodds TJ, Patch AM, Nones K, Tembe V, Shang P, van der Weyden L, Wong K, Holmes O, Lo S, Leonard C, Wood S, Xu Q, Rawson RV, Mukhopadhyay P, Dummer R, Levesque MP, Jonsson G, Wang X, Yeh I, Wu H, Joseph N, Bastian BC, Long GV, Spillane AJ, Shannon KF, Thompson JF, Saw RPM, Adams DJ, Si L, Pearson JV, Hayward NK, Waddell N, Mann GJ, Guo J, Scolyer RA. Whole-genome landscape of mucosal melanoma reveals diverse drivers and therapeutic targets. Nat Commun. 2019 Jul 18;10(1):3163. doi: 10.1038/s41467-019-11107-x. PMID 31320640
- [Result] Sheen YS, Tan KT, Tse KP, Liao YH, Lin MH, Chen JS, Liau JY, Tseng YJ, Lee CH, Hong CH, Liao JB, Chang HT, Chu CY. Genetic alterations in primary melanoma in Taiwan. Br J Dermatol. 2020 May;182(5):1205-1213. doi: 10.1111/bjd.18425. Epub 2019 Oct 15. PMID 31408190
- [Result] Chang JW, Guo J, Hung CY, Lu S, Shin SJ, Quek R, Ying A, Ho GF, Nguyen HS, Dhabhar B, Sriuranpong V, Tiambeng ML, Prayogo N, Yamazaki N. Sunrise in melanoma management: Time to focus on melanoma burden in Asia. Asia Pac J Clin Oncol. 2017 Dec;13(6):423-427. doi: 10.1111/ajco.12670. Epub 2017 Feb 15. No abstract available. PMID 28198155
- [Result] Wu CE, Yang CK, Peng MT, Huang PW, Lin YF, Cheng CY, Chang YY, Chen HW, Hsieh JJ, Chang JW. Immune Checkpoint Inhibitors for Advanced Melanoma: Experience at a Single Institution in Taiwan. Front Oncol. 2020 Jun 4;10:905. doi: 10.3389/fonc.2020.00905. eCollection 2020. PMID 32582554